CLINICAL TRIAL: NCT02091895
Title: Validation of Clinical Efficacy and Development of New Diagnostic Algorithm of Probe-based Confocal Laser Endomicroscopy in Patients With Lower Gastrointestinal Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2013-0942
Record Dates: First submitted 2014-03-16; First posted 2014-03-19 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Lower Gastrointestinal Disorders
Keywords: probe-based confocal laser endomicroscopy, lower gastrointestinal disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endo group (Experimental): colon polyp, early colon cancer, colorectal submucosal tumor, ileocecal ulcers
  Interventions: Procedure: probe-based confocal laser endomicroscopy

INTERVENTIONS:
Procedure: probe-based confocal laser endomicroscopy — After shooting 10% fluorescein sodium in,2.5-5 .0 ml to the object with colorectal disease, the lesion will observed and evaluated with pCLE in real-time and also stored the inspection images.
  Then, determines the treatment plan to determine which is applied currently in clinical, Sensitivity, specificity, accuracy, amphoteric predict of pCLE diagnosis, and calculate the agreement of prediction compared to the pathological findings of lesions Based on the inspection image stored, using Delphi approach tests, two or more are discussed, to derive a significant technical phrases.
  Check diagnostic agreement of technical phrases which are derived, the matching degree between observers, and developed a new classification method based on this.

SUMMARY:
The aims of this research are to validate and develop of therapeutic strategies for patients with colorectal lesions in real time through pCLE(probe-based confocal laser endomicroscopy). Endomicroscopy is a technique for obtaining histology-like images from inside the human body in real-time. Total objections are 311 patients.

Specific research topics are as below.

1. Diagnosis and classification of colon polyps through pCLE
2. Evaluation of the depth of invasion of colorectal cancer or lateral growth type tumor through the pCLE
3. Differential diagnosis of colorectal submucosal tumor through the pCLE
4. Differential diagnosis of ileocecal ulcers through the pCLE

The study will be conducted to measure sensitivity, specificity, accuracy, amphoteric predict of pCLE diagnosis, and calculate the agreement of prediction compared to the pathological findings of lesions Check diagnostic agreement of technical phrases which are derived, the matching degree between observers, and will develope a new classification method based on this.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years old
* Patients with colorectal polyps
* Patients who undergo endoscopic submucosal dissection (ESD) due to lateral spreading tumors or early colorectal cancer
* Patients with submucosal tumor in colorectal cancer
* Patients with ileocecal ulcers
* Patients who consented to research

Exclusion Criteria:

* Patients who are impossible to biopsy or polypectomy due to underlying diseases.
* Patients who are not able to end the ESD because of a complication
* Patients who are already known the cause of ileocecal ulcers before the pCLE.
* Patients with contraindications to the use of disease fluorescent contrast agents
* Patients who did not consent to research
* Patients who are unsuitable for clinical trials in charge of the attending physician.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Estimated)
Dates: Start 2014-03; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of pCLE diagnosis | 2 weeks
  The study will be conducted to measure sensitivity, specificity, accuracy, amphoteric predict of pCLE diagnosis, and calculate the agreement of prediction compared to the pathological findings of lesions.

SECONDARY OUTCOMES:
Specificity of pCLE diagnosis | 2 weeks
  The study will be conducted to measure sensitivity, specificity, accuracy, amphoteric predict of pCLE diagnosis, and calculate the agreement of prediction compared to the pathological findings of lesions.
Accuracy of pCLE diagnosis | 2 weeks
  The study will be conducted to measure sensitivity, specificity, accuracy, amphoteric predict of pCLE diagnosis, and calculate the agreement of prediction compared to the pathological findings of lesions.
amphoteric predict of pCLE diagnosis | 2 weeks
  The study will be conducted to measure sensitivity, specificity, accuracy, amphoteric predict of pCLE diagnosis, and calculate the agreement of prediction compared to the pathological findings of lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea